CLINICAL TRIAL: NCT05467852
Title: Didroxyprogesterone Promotes Postoperative Natural Pregnancy in Infertile Patients With Mild and Moderate Endometriosis
Brief Title: Didroxyprogesterone Promotes Natural Pregnancy in Infertile Patients With Endometriosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Shenzhen People's Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-026
Record Dates: First submitted 2022-04-01; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy Rate
MeSH Terms: interventions — Dydrogesterone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Didroxyprogesterone treatment group (Active Comparator): Since the first menstrual cycle after surgery, dydrogesterone was administered orally 10mg bid on the 14th to 27th day of each menstrual cycle, planned to be used for 6 menstrual cycles (if the patient conceived naturally during medication, the drug could be stopped), and the patient was instructed to try pregnancy, the observation period was 12 menstrual cycles after surgery.
  Interventions: Drug: didroxyprogesterone
- control (No Intervention): No medication was used after surgery, and the observation period was 12 menstrual cycles after surgery

INTERVENTIONS:
Drug: didroxyprogesterone — Didroxyprogesterone group: the first menstrual cycle after operation began on the 14th to 27th day of each menstrual cycle. Didroxyprogesterone 10mg bid was given orally. It was planned to use 6 menstrual cycles (if the patient was naturally pregnant during the medication, the drug could be stopped), and guide the patient to try pregnancy. The observation period was 12 menstrual cycles after operation. Control group: no drugs were used after operation, and the patients were guided to try pregnancy. The observation period was 12 menstrual cycles after operation. Subjects need to complete up to 6 follow-up visits, including the first month after operation, the first menstrual cycle d7-13 after operation, the fourth menstrual cycle d7-13 after operation, the seventh menstrual cycle d7-13 after operation, the 13th menstrual cycle d7-13 after operation and 1-2 months after termination of pregnancy
  Other Names: duphaston
  Arms: Didroxyprogesterone treatment group

SUMMARY:
Endometriosis (EM) is an important cause of infertility in women of childbearing age. Laparoscopic surgery is the treatment of EM Related infertility is an important method. However, excluding other infertility factors, the natural pregnancy rate of EM patients one year after operation is still significantly lower than that of normal couples. At the same time, the high recurrence rate of EM often requires drugs to inhibit ovulation after operation, which forms a paradox with the demand for fertility. One year after operation is the "golden period" of natural pregnancy. Whether to treat the recurrence of EM without affecting or even promoting fertility is a key problem to be solved in clinic. Didroxyprogesterone is the closest natural progesterone. It is widely used in luteal support and treatment of threatened abortion. It does not affect ovulation and is harmless to embryos. In recent years, clinical studies have found that it is helpful to the natural pregnancy of patients with EM after operation, and is beneficial to improve pain symptoms and reduce the recurrence rate. Basic studies have also confirmed the inhibitory effect of didroxyprogesterone on em. However, the existing studies with small sample size are not enough to draw a convincing conclusion that didroxyprogesterone promotes the pregnancy rate after em, and there is a lack of Chinese data. This study intends to use a multicenter, prospective, open, randomized controlled clinical trial design to explore the value of didroxyprogesterone in the treatment of EM related infertility patients, so as to provide direct evidence for improving the postoperative natural pregnancy rate of EM patients.

DETAILED DESCRIPTION:
Female patients aged 22-35 who had been diagnosed with mild to moderate endometriosis by laparoscopic surgery and had undergone surgical treatment and fertility index (EFI) score ≥5 were stratified and randomized at each branch center. The study subjects were first stratified according to EFI score, which was divided into three levels: 5-6 points, 7-8 points and 9-10 points. Then the patients were divided into 2 groups in stratification according to the segmented random method. ① Dydrogesterone group: the first postoperative menstrual cycle began on the 14th to 27th day of each menstrual cycle, dydrogesterone 10mg bid oral administration, planned to use 6 menstrual cycles (if the patient conceived naturally during the medication, the drug could be stopped), and instructed the patient to try pregnancy, observation period was 12 postoperative menstrual cycles; ② Control group: postoperative medication was not used to guide patients to try pregnancy, and the observation period was 12 menstrual cycles after surgery. The subjects should be followed up for a maximum of 6 times, respectively within the first month after surgery, the first menstrual cycle D7-13 after surgery, the fourth menstrual cycle D7-13 after surgery, the seventh menstrual cycle D7-13 after surgery, the 13th menstrual cycle D7-13 after surgery, and 1-2 months after pregnancy termination.

Outcome measures: ① Pregnancy status; ②EM symptoms and recurrence related indicators: VAS score, physical examination, CA125, gynecological B-ultrasound examination results; ③ Drug safety assessment: AMH, blood routine examination, liver and kidney function, and the patient's combined drug use and possible drug-related adverse reactions were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 22 years and ≤ 35 years, diagnosed as infertility and with reproductive needs;
* BMI：18.5-27.9kg/m2；
* The menstrual cycle in recent half a year is 21-35 days;
* Laparoscopic surgery was performed in certain hospitals, the intraoperative diagnosis or postoperative pathological diagnosis was em, and the EM fertility index (EFI) score was ≥ 5; .Patients agreed to conduct the study and signed informed consent.

Exclusion Criteria:

* There are contraindications to the use of didroxyprogesterone;
* Vaginal rectal septum, endometrial em, recurrent em;
* The ovarian reserve function decreased after operation, AMH < 1.1 ng / ml or premature ovarian failure;
* Unilateral or bilateral tubal obstruction or effusion;
* Combined uterine diseases: uterine malformation (single horn uterus, double horn uterus, double uterus, mediastinal uterus); Combined with adenomyosis and intrauterine adhesion;
* Chromosomal abnormalities of both husband and wife or one of them;
* Men with abnormal semen analysis results, low spermatogenic function, non obstructive azoospermia or AZF gene microdeletion; .patients with contraindications of pregnancy: uncontrolled diabetes, undiagnosed liver and kidney dysfunction, deep venous thrombosis, history of pulmonary embolism, history of cerebrovascular accident, uncontrolled hypertension, heart disease, suspicious cervical cancer, endometrial cancer, history of breast cancer or previous history, and undiagnosed vaginal bleeding;. No long-term follow-up or poor compliance, or the investigator believes that there are any factors that affect the subject's participation in the trial or result evaluation.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 6 weeks
  percentage

IPD SHARING:
Plan to Share IPD: No